CLINICAL TRIAL: NCT01915069
Title: Cilostazol and Its Effects on Human Oocyte Maturation in Vivo: A Pilot Study
Brief Title: Cilostazol and Its Effects on Resumption of Meiosis in the Human Ovary
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Laura Sech, Family Planning Research Fellow, Department OBGYN, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SFPRF 13-14
Record Dates: First submitted 2013-07-05; First posted 2013-08-02 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Contraception
Keywords: contraception; Cilostazol; phosphodiesterase inhibitors; To assess the ability of Cilostazol to act as a contraceptive agent
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cilostazol (Experimental): The primary aim of the study is to assess the affects of oral Cilostazol taken at the FDA approved dose of 100mg PO bid on human oocyte maturation.
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Cilostazol
  Other Names: Pletal

SUMMARY:
Combined oral contraceptive pills (COCs) are the most commonly used hormonal form of birth control in the United States with at least 87% of women of reproductive age reporting oral contraceptive use at some point in their lives (9). Despite their frequent use, the six and twelve month discontinuation rates for oral contraceptive pills are 31 and 47 % respectively (17), with common reasons for discontinuation attributed to the side effects of abnormal bleeding, headache, and weight gain.

Additionally, COCs are contraindicated in certain groups of women as outlined by The Centers for Disease Control Medical Eligibility Criteria (11). Given the high prevalence of oral contraceptive users who commonly discontinue use secondary to side effects or who are not eligible for use as a result of underlying health conditions, the development of novel oral non-hormonal methods that are equally effective at pregnancy prevention are warranted.

This current study aims to evaluate the effect of an FDA approved drug, Cilostazol, on human oocyte maturation. Such a study has not been conducted to date. If Cilostazol demonstrates an ability in humans to affect resumption of meiosis, then this non-hormonal agent could be uses as a possible contraceptive agent in the future. This knowledge would have profound reproductive health implications.

The investigators propose that women undergoing treatment with the FDA approved dose of 100mg PO every 12 hours of Cilostazol will demonstrate an impairment of egg maturation in comparison to paired historic controls following ovarian follicle stimulation.

DETAILED DESCRIPTION:
Combined oral contraceptive pills (COCs) are the most commonly used hormonal form of birth control in the United States with at least 87% of women of reproductive age reporting oral contraceptive use at some point in their lives (9). Despite their frequent use, the six and twelve month discontinuation rates for oral contraceptive pills are 31 and 47 % respectively (17), with common reasons for discontinuation attributed to the side effects of abnormal bleeding, headache, and weight gain.

Additionally, COCs are contraindicated in certain groups of women as outlined by The Centers for Disease Control Medical Eligibility Criteria (11). Given the high prevalence of oral contraceptive users who commonly discontinue use secondary to side effects or who are not eligible for use as a result of underlying health conditions, the development of novel oral non-hormonal methods that are equally effective at pregnancy prevention are warranted.

The potential for the development of non-hormonal contraception has been present in the scientific literature since the 1980s at which point the critical components of gametogenesis of the mammalian oocyte were being classified. Bornslaeger and colleagues discovered that high concentrations of intracellular cAMP, an important second messenger for many biological processes, inhibited resumption of meiosis I in mouse oocytes (3). Later studies demonstrated that phosphodiesterase 3 inhibitors, capable of preventing the breakdown of cAMP, were able to prevent resumption of meiosis in mouse oocytes cultured in vitro (6).

Since the 1980s, additional studies have examined phosphodiesterase inhibitors and their role in prevention of oocyte maturation. Tsafriri and colleagues showed that phosphodiesterase inhibitors were able to exert their effects selectively via type specific isoforms. This study revealed that granulosa cells exert effects via type 4 phosphodiesterase inhibitors and oocytes respond to signals via type 3 phosphodiesterase inhibitors such that oocyte maturation was prevented in the presence of PDE3 inhibitors yet ovulation was unaffected (15). Most recently, Jensen and colleagues examined both in vitro and in vivo effects of a phosphodiesterase 3 inhibitor ORG 9935 on oocyte maturation in rhesus monkeys. In these animal studies, it was found that in vitro, ORG 9935 at a concentration of 1.0umol/l was able to completely inhibit oocyte maturation (7).

In vivo models demonstrated a similar reduction in oocyte maturation, with the most dramatic reduction in monkeys treated with an extended dose regimen of ORG 9935 (200mg/kg/d) prior to ovulation (8). Additionally, pregnancy rates in macaques treated with ORG 9935 was studied and compared to controls. Overall, there was not a statistically significant decrease in pregnancy rates in those macaques treated with PDE3 inhibitor; however, there did appear to be evidence of a dose response as no animal became pregnant who had serum ORG 9935 levels above 300nM/L (9). Despite a clear dose response, authors of this study acknowledge that PDE3-Is have systemic effects that are also dose-limiting. At higher doses, adverse effects such as tachycardia and hypotension were observed.

Phosphodiesterase 3 inhibitors have additionally been studied in vitro to assess oocyte maturation in humans. Human oocytes cultured in the presence of ORG 9935 (1um) for 24 hours demonstrated a statistically significant reduction in germinal vesicle breakdown (an early marker of oocyte maturation) in comparison to control oocytes (12). However, no human in vivo models assessing oocyte maturation following treatment with a phosphodiesterase 3 inhibitor exist.

Cilostazol, an FDA approved drug for the treatment of intermittent claudication, is a class IIIa phosphodiesterase inhibitor. Its systemic effects in humans include vasodilation, decrease in platelet aggregation, reduction in triglyceride levels, and increase in HDL cholesterol levels (4). Human clinical trials did not address fertility and pregnancy rates; however, manufacturer product labeling reports that no fertility effects occurred in rats. Most recently, however, two animal in vivo studies examining pregnancy rates of mice treated with Cilostazol were conducted (1,10). In both of these studies, mice treated with Cilostazol were shown to be completely infertile at follow up; however, once the drug was discontinued, all mice that were unable to conceive during treatment with cilostazol were subsequently able to have pregnancies of normal litter sizes. It is important to mention that in the study by Albarzanchi, mice received PO cilostazol at a dose of 7.5 or 15 mg PO for three days (1). In the study by Li conducted in China, the maxium dose was higher (300mg/kg) (10). Pregnancy outcomes for both studies were the same.

These studies demonstrate two important aspects of a contraceptive method: efficacy and reversibility. Additionally, the investigators who published Cilostazol's fertility effects in mice published an abstract demonstrating a similar effect in swine (2). When a human dose of 100mg bid of Cilostazol was given prior to ovulation, no documented pregnancies occurred. Following cessation of study drug, all swine were able to conceive.

Given the success of phosphodiesterase inhibitors in both in vivo and in vitro models for prevention of oocyte maturation and pregnancy in animal models, it is reasonable that we further examine this potential non-hormonal oral contraceptive method. Given the many FDA clinical trials that need to be conducted, new contraceptive methods take decades to develop. However, since Cilostazol is an approved FDA medication with an acceptable side effect profile, we believe that it is appropriate to complete initial studies of this drug in humans using an in vivo technique validated in macaques, a model with the same timing of peri-ovulatory events as women, to ascertain its possible use as a non-hormonal oral contraceptive.

The primary objective of the research study is to determine if women taking Cilostazol demonstrate impairment of oocyte maturation in comparison to paired historic controls following ovarian follicle stimulation. For the purposes of our study, oocyte maturation will be assessed using the oocyte maturational stages of prophase I, metaphase I, and metaphase II. Thus, we will be assessing the percent of oocytes aspirated from follicles during controlled ovarian stimulation that progress beyond the germinal vesicle stage (e.g. GVBD) in those women receiving cilostazol and compare this to the maturation of oocytes obtained from the same women who underwent ovarian follicle stimulation previously while not on study drug.

We propose that women undergoing treatment with the FDA approved dose of 100mg PO BID of Cilostazol will demonstrate an impairment of oocyte maturation in comparison to paired historic controls following ovarian follicle stimulation.

ELIGIBILITY:
Inclusion Criteria:

* previous oocyte donor in USC IVF clinic within past 3 years
* age 18-33
* willingness and ability to commit to the time requirements of the study
* willingness to donate oocytes for research purposes
* willingness to discontinue current hormonal contraception
* otherwise healthy subjects

Exclusion Criteria:

* contraindications to combined hormonal contraceptive use (CDC MEC class 3 or 4)
* pregnancy
* history of cardiac arrhythmias
* history of heart failure
* history of bleeding disorder
* concomitant use of anti-platelet therapy such as aspirin
* current use of drugs that inhibit cytochrome P450 CYP 3A4 (erythromycin, diltiazem, ketoconazole, itraconazole) or CYP 2C19 (omeprazole) as they may lead to increased serum levels of cilostazol.

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Oocyte maturation | 6 weeks
  For the purposes of our study, oocyte maturation will be assessed using the oocyte maturational stages of prophase I, metaphase I, and metaphase II. Thus, we will be assessing the percent of oocytes aspirated from follicles during controlled ovarian stimulation that progress beyond the germinal vesicle stage (e.g. GVBD) in those women receiving cilostazol and compare this to the maturation of oocytes obtained from the same women who underwent ovarian follicle stimulation previously while not on study drug.

OTHER OUTCOMES:
Serum and follicular fluid cilostazol levels | 6 weeks
  Serum and follicular fluid cilostazol levels will be collected for each participant throughout the treatment phase to ensure adherence to medication and to correlate cilostazol levels to degree of oocyte maturation at the time of egg retrieval.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California Fertility Clinic, Los Angeles, California, United States